CLINICAL TRIAL: NCT00301951
Title: Pilot Study of Reduced-Intensity Umbilical Cord Blood Transplantation in Adult Patients With Advanced Hematopoietic Malignancies
Brief Title: Low-Dose Fludarabine, Busulfan, and Anti-Thymocyte Globulin Followed By Donor Umbilical Cord Blood Transplant in Treating Patients With Advanced Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000465362; UCSF-04253; UCSF-2407; UCSF-H24045-25271-02
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; angioimmunoblastic T-cell lymphoma; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; anaplastic large cell lymphoma; nodal marginal zone B-cell lymphoma; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; refractory chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage IV adult T-cell leukemia/lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III small lymphocytic lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Immunoblastic Lymphadenopathy; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Antilymphocyte Serum; sargramostim; Busulfan; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- cord blood transplant (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: sargramostim; Drug: busulfan; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: sargramostim
Drug: busulfan
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor umbilical cord blood transplant helps stop both the growth of cancer cells and the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving chemotherapy, such as fludarabine and busulfan, and antithymocyte globulin before transplant and tacrolimus and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This clinical trial is studying how well giving low-dose fludarabine and busulfan together with anti-thymocyte globulin, followed by donor umbilical cord blood transplant works in treating patients with advanced hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the feasibility of performing umbilical cord blood transplants in older patients or younger infirm patients with advanced hematologic malignancies using a reduced-intensity preparative regimen, as determined by > 80% engraftment rate at day 180 and a < 50% transplant-related mortality rate at day 100.

Secondary

* Describe the time to neutrophil and platelet recovery in patients treated with this regimen.
* Determine disease-specific, event-free, and overall survival rate at days 180 and 360.
* Determine the incidence, severity, and timing of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Evaluate T-cell, B-cell, and natural killer cell recovery in patients treated with this regimen.
* Assess lineage-specific chimerism after transplantation and describe the contribution of each individual cord blood unit to post-transplantation hematopoiesis.

OUTLINE: This is a pilot study.

* Reduced-intensity preparative regimen: Patients receive fludarabine IV over 30 minutes on days -8 to -4, busulfan IV over 2 hours 4 times daily on days -4 and -3, and anti-thymocyte globulin IV over 6 hours on days -3 to -1.
* Allogeneic umbilical cord blood transplantation: Patients undergo allogeneic umbilical cord blood transplant on day 0. Patients receive sargramostim (GM-CSF) subcutaneously or IV beginning on day 7 and continuing until blood counts recover.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive tacrolimus IV continuously over 24 hours or orally (as tolerated) beginning on day -2 and continuing for approximately 9 months. Patients also receive oral mycophenolate mofetil twice daily on days 1-50.

After completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following advanced hematologic malignancies:

  * Acute myeloid leukemia (AML) meeting the following criteria:

    * Considered incurable with chemotherapy
    * Marrow blasts ≤ 10% (may be achieved using standard chemotherapy regimen)
    * Meets any of the following criteria:

      * High-risk cytogenetics (-7, -7q, -5, -5q, t(6,9), t(9,11), complex [≥ 3 abnormalities], Philadelphia chromosome positive [Ph+])
      * AML evolved from prior myelodysplasia
      * AML secondary to prior chemotherapy
      * Failed to achieve remission
      * In second or subsequent remission
      * Refractory relapse
  * Myelodysplastic syndromes (MDS) meeting the following criteria:

    * Must have high-risk features, including any of the following:

      * Intermediate-2 or high risk International Prognostic Scoring System (IPSS) score
      * Chronic myelomonocytic leukemia
    * Marrow blasts ≤ 20% (chemotherapy may be given to achieve target blast levels)
    * No rapidly progressive disease
  * Acute lymphoblastic leukemia meeting the following criteria:

    * Considered incurable with chemotherapy
    * Meets any of the following criteria:

      * High-risk cytogenetics (Ph+, t(4,11), 11q23 abnormalities, or monosomy 7)
      * Required > 1 induction course to achieve remission
      * Failed to enter remission
      * In second or subsequent remission
    * Marrow blasts ≤ 10% (chemotherapy may be given to achieve target blast levels)
  * Chronic myelogenous leukemia (CML) meeting 1 of the following criteria:

    * Chronic phase CML that failed imatinib mesylate therapy, as defined by progressive disease or failed to achieve a major cytogenetic response at 1 year after initiation of therapy
    * Accelerated phase CML meeting 1 of the following criteria:

      * Failed to achieve a complete cytogenetic remission at 1 year after initiation of therapy
      * Failed to achieve any cytogenetic response after 6 months of therapy
      * Progressive disease, as demonstrated by worsening cytogenetic response in 2 consecutive analyses separated by 4 weeks
    * In blast crisis with < 10% blasts in bone marrow
  * Multiple myeloma meeting the following criteria:

    * Stage I-III disease
    * Meets any of the following criteria:

      * In relapse after autologous transplantation
      * Refractory to ≥ 2 prior conventional myeloma therapies
      * Chromosome 13 abnormalities (may be enrolled at diagnosis or after initial progression)
  * Lymphoma

    * The following subtypes are eligible:

      * Diffuse large cell
      * Follicular large cell
      * Mantle cell
      * Peripheral T-cell
      * T-natural killer (T-NK) cell
      * Hodgkin's lymphoma
    * Must have progressed, recurred after prior therapy, or failed to respond to primary therapy
    * Relapsed disease after autologous stem cell transplantation (SCT) allowed
  * Low-grade non-Hodgkin's lymphoma meeting 1 of the following criteria:

    * Relapsed or refractory disease after ≥ 2 chemotherapy-based treatment regimens
    * Relapsed after autologous SCT
  * Chronic lymphocytic leukemia

    * Relapsed or refractory disease after ≥ 2 chemotherapy-based treatment regimens
    * Relapsed after autologous SCT
* Meets 1 of the following criteria:

  * Age 55-70 years
  * Under age 55 and deemed ineligible for conventional high-dose chemotherapy, as indicated by any of the following:

    * Poor cardiac function (i.e., LVEF < 40%)
    * Poor pulmonary function (i.e., DLCO < 50%)
    * Hepatic dysfunction
    * Prior myeloablative therapy
* Not eligible for autologous SCT or conventional therapy
* Umbilical cord blood donor available

  * Matched at ≥ 4 of 6 HLA antigens (A, B, and DR)
  * Has 1-3 units of umbilical cord blood available
  * Must not have an HLA-identical or 1 antigen mismatched related donor or potential HLA-matched unrelated donor readily available NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine clearance > 40 mL/min
* Creatinine < 2.0 mg/dL
* AST and alkaline phosphatase < 3 times upper limit of normal (ULN)
* Bilirubin < 2.0 mg/dL
* Hepatitis C or active hepatitis B virus (HBV) allowed if ≤ grade 2 fibrosis and/or inflammation by liver biopsy

  * Patients with history of HBV infection should be tested for hepatitis B epsilon (HBe) antigen, anti-HBe, and HBV DNA (quantitative)
  * Patients with active HBV viral replication should receive antiviral therapy
* Ejection fraction > 30%
* DLCO ≥ 40%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring ongoing antibiotic treatment
* HIV negative

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility of donor cord blood transplant | up to 36 months post transplant
  as determined by > 80% engraftment rate at day 180 and a < 50% transplant-related mortality rate at day 100

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States